CLINICAL TRIAL: NCT01007526
Title: Open-labeled, Multicenter Phase II Study of Concomitant Chemo-radiotherapy Followed by VIDL Chemotherapy With Risk-based Application of Autologous Stem Cell Transplantation in Stage I/II Extranodal NK/T-cell Lymphoma
Brief Title: Concomitant Chemo-radiotherapy Plus VIDL Chemotherapy in NK/T-cell Lymphoma
Acronym: CCRT-VIDL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); National Cancer Center, Korea (Other Government); Severance Hospital (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-04-033
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-09

CONDITIONS: NK/T-cell Lymphoma of Nasal Cavity
Keywords: Extranodal Lymphoma; Natural killer cell; T cell; Radiotherapy; Chemotherapy

STUDY DESIGN:
Intervention Model Description: VIDL (Etoposide, ifosfamide, dexamethasone and L-asparaginase)
Masking Description: Concomitant Chemo-radiotherapy Plus VIDL Chemotherapy
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCRT plus VIDL (Experimental): CCRT followed by VIDL chemotherapy Concomitant chemo-radiotherapy followed by VIDL chemotherapy with risk-based application of autologous stem cell transplantation Patients who are planned to be treated with CCRT plus VIDL chemotherapy and/or autologous stem cell transplantation
  Interventions: Other: CCRT followed by VIDL chemotherapy

INTERVENTIONS:
Other: CCRT followed by VIDL chemotherapy — CCRT followed by VIDL chemotherapy concomitant chemo-radiotherapy followed by VIDL (VP-16, Ifosfamide, Dexamethasone, L-asparaginase) chemotherapy with risk-based application of autologous stem cell transplantation

SUMMARY:
This study is to evaluate the efficacy of risk-adapted treatment strategy for stage I/II extranodal NK/T cell lymphoma. The risk stratification is based on the Korean NK prognostic index. Thus, the group I/II will receive concomitant chemoradiation followed by VIDL chemotherapy. The group III/IV will receive high dose-chemotherapy followed by autologous stem cell transplantation after the completion of VIDL chemotherapy.

DETAILED DESCRIPTION:
1. Concomitant chemo-radiotherapy:

   Radiotherapy 36-44 Gy/18-22 fractions

   + weekly cisplatin 30 mg/m2 for 4 weeks
2. Rest period: 3 weeks
3. VIDL combination chemotherapy: (total 2 cycles) VP-16 (etoposide) 100mg/m2 I.V. D1-3 Ifosfamide 1.2g/m2 I.V. D1-3 Dexamethasone 40mg/day D1-3 L-asparaginase 4000IU/m2 IM D8, 10, 12, 14, 16, 18, 20 Repeated every 28 days
4. Peripheral blood stem cell mobilization G-CSF 400ug/m2/day or 10ug/kg/day S.C. or I.V. for 4-6 days followed by stem cell collection (Minimum requirement of CD34+ cells > 2×106/kg)
5. High-dose chemotherapy with autologous stem cell transplantation Busulfex 3.2mg/kg/day from day -7 to day -5 Etoposide 400mg/m2/day on day -5, -4 Cyclophosphamide 50mg/kg/day on day -3, -2 Followed by stem cell infusion

ELIGIBILITY:
Inclusion Criteria:

* patients were required to have a biopsy-proven diagnosis of nasal ENKTL
* at least 18 years old
* Ann Arbor stage IE or IIE
* measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* life expectancy greater than 12 weeks
* adequate hematologic (hemoglobin > 9.0 g/dL, absolute neutrophil count > 1,500/uL and platelets > 100,000/uL)
* renal (serum creatinine < 1.5 mg/dL, creatinine clearance > 50 mL/min)
* hepatic (total bilirubin < 2 times of upper limit of normal and aspartate transferase < 3 times of upper limit of normal) function
* Diagnosis of ENKTL is based on the presence of histological features and immunophenotypes compatible with ENKTL (e.g., cytoplasmic CD3+, CD20-, CD56+, positive for cytotoxic molecules, positive for EBV by in situ hybridization).
* Informed consent

Exclusion Criteria:

* prior or concomitant malignant tumors
* any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol.
* ENKTL with non-nasal sites such as skin or gastrointestinal tract was excluded even if it is localized.
* Other subtypes of non-Hodgkin lymphoma (NHL), including myeloid/NK cell precursor acute leukemia, blastic NK cell lymphoma/precursor NK cell lymphoblastic leukemia, aggressive NK cell leukemia, and peripheral T cell lymphoma, unspecified, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between August 2008 and October 2010 Location: University hospital or Institutes
Period: Overall Study
Arm/Group | CCRT Plus VIDL
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CCRT Plus VIDL
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 31

OUTCOME MEASURES:

1. Primary Outcome: Compete Response Rate
Description: Response was determined by the revised response criteria for malignant lymphoma (Cheson BD et al. J Clin Oncol. 2007 Feb 10;25(5):579-86.): 1) Complete response 2) Partial response 3) Stable disease 4) Progressive disease
Time Frame: Within 3 weeks after the completion fo treatment
Measure: Number; unit: participants
Arm/Group | CCRT Plus VIDL
Number analyzed (Participants) | 31
participants | 31

2. Secondary Outcome: Overall Response Rate, Survival, Toxicity
Time Frame: Up to 5 years after the completion of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months after registration
Description: We applied the same definition as the clinicaltrials.gov.
Arm/Group | CCRT Plus VIDL
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCRT Plus VIDL (N=30)
Neutropenia (Blood and lymphatic system disorders) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes